CLINICAL TRIAL: NCT00278447
Title: Linkage of Alcohol Abusers to Primary Care
Brief Title: Addiction Health Evaluation And Disease Management (AHEAD) Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SAI-010870-06A2; P60AA013759 (NIH); NIAAA Grant 2R01 AA010870-06A2; NIDA Grant 2R01 DA010019-07A1
Record Dates: First submitted 2006-01-13; First posted 2006-01-18 (Estimated); Last update posted 2014-10-02 (Estimated); Status verified 2012-10

CONDITIONS: Alcohol Dependence; Alcoholism; Drug Dependence
Keywords: Alcohol; Alcohol use; Alcohol dependence; Drug; Drug use; Drug dependence; Utilization; Hospitalization; Primary care; Chronic disease management; Care management; Comorbidity
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders; Alcohol Drinking; Patient Acceptance of Health Care | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1) CDM (Active Comparator): Chronic Disease Management
  Interventions: Behavioral: Chronic Disease Management for substance abuse
- 2) Standard care (Active Comparator): Standard care
  Interventions: Behavioral: Standard care

INTERVENTIONS:
Behavioral: Chronic Disease Management for substance abuse — Referral to primary medical care & longitudinal, multidisciplinary care for persons with substance dependence.
  Arms: 1) CDM
Behavioral: Standard care — Referral to primary medical care for persons with substance dependence.
  Arms: 2) Standard care

SUMMARY:
The objective of this study is to test whether a chronic disease management (CDM) program for substance abusers in primary care leads to improved alcohol and drug-related outcomes (such as reduced consumption and health problems) and health care utilization patterns.

DETAILED DESCRIPTION:
Chronic disease management (CDM) is a collaborative, longitudinal, proven effective approach to the treatment of chronic medical illnesses that addresses individual patient and health systems barriers to receipt of needed treatment. The objective of this Addiction Health Evaluation And Disease management (AHEAD) Study is to test the effectiveness of CDM for substance dependence in primary care. The study will enroll and randomize subjects to attend a substance dependence CDM program (the AHEAD Unit) integrated into a real-world primary care clinic or to referral to usual primary care. All subjects will be assessed regarding alcohol and/or drug diagnosis, consumption and problems, readiness to change, health-related quality of life, and medical and substance abuse treatment utilization. Primary outcomes are alcohol and drug use, alcohol and drug-related problems, emergency department visits, and hospitalizations. Additional outcomes are health-related quality of life, readiness to change, medical and psychiatric comorbidity, HIV risk behaviors, and treatment utilization and costs. The hypothesis is that compared with standard care, a health services intervention -- chronic disease management for alcohol and drug dependence integrated in primary care -- will decrease alcohol and drug use and related problems, and improve health care utilization patterns.

This study contains two studies (and study populations):

* 1. 320 alcohol dependent subjects with current risky drinking, and
* 2. 320 drug dependent subjects with current drug use.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Fluent in English or Spanish
* Alcohol or drug dependent
* Heavy drinking in the past 30 days or recent drug use
* Provide 2 contacts to assist with follow-up
* Have no plans to move from the local area within a year of screening
* Score >21 on Mini-Mental State Examination (no serious cognitive impairment)

Exclusion Criteria:

* Pregnant (self-report)
* Breath alcohol >100 mg/dL
* Inability to provide informed consent determined by trained research associates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2006-04; Primary Completion 2010-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Alcohol and drug use | 3, 6, and 12 months after baseline
Alcohol and drug-related problems | 3, 6, and 12 months after baseline
Nights Hospitalized | 3, 6, and 12 months after baseline and up to 2 years after the last subject is enrolled
Emergency department visits | 3, 6, and 12 months after baseline and up to 2 years after the last subject is enrolled

SECONDARY OUTCOMES:
Health-related quality of life | 3, 6, and 12 months after baseline
Readiness to change | 3, 6, and 12 months after baseline
Medical comorbidity | 3, 6, and 12 months after baseline
Psychiatric comorbidity | 3, 6, and 12 months after baseline
HIV risk behaviors | 3, 6, and 12 months after baseline
Treatment utilization and costs | 3, 6, and 12 months after baseline, and up to 2 years after the last subject is enrolled

CONTACTS AND LOCATIONS:
Overall Officials: Richard Saitz, MD, MPH, Principal Investigator — Boston University
Locations (1):
- Boston Medical Center / Boston University, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Park TW, Samet JH, Cheng DM, Winter MR, Kim TW, Fitzgerald A, Saitz R. The prescription of addiction medications after implementation of chronic care management for substance dependence in primary care. J Subst Abuse Treat. 2015 May;52:17-23. doi: 10.1016/j.jsat.2014.11.008. Epub 2014 Dec 2. PMID 25524751
- [Derived] Park TW, Cheng DM, Samet JH, Winter MR, Saitz R. Chronic care management for substance dependence in primary care among patients with co-occurring disorders. Psychiatr Serv. 2015 Jan 1;66(1):72-9. doi: 10.1176/appi.ps.201300414. Epub 2014 Nov 17. PMID 25219686
- [Derived] Saitz R, Cheng DM, Winter M, Kim TW, Meli SM, Allensworth-Davies D, Lloyd-Travaglini CA, Samet JH. Chronic care management for dependence on alcohol and other drugs: the AHEAD randomized trial. JAMA. 2013 Sep 18;310(11):1156-67. doi: 10.1001/jama.2013.277609. PMID 24045740
- [Derived] D'Amore MM, Cheng DM, Allensworth-Davies D, Samet JH, Saitz R. Disparities in safe sex counseling & behavior among individuals with substance dependence: a cross-sectional study. Reprod Health. 2012 Dec 31;9:35. doi: 10.1186/1742-4755-9-35. PMID 23276300